CLINICAL TRIAL: NCT07324564
Title: A Randomized, Evaluator-blinded, No-treatment Controlled, Multicenter Study to Evaluate the Effectiveness and Safety of Sculptra 011611 for Improvement in Appearance of Gluteal Skin Irregularities
Brief Title: Safety and Effectiveness of Sculptra 011611 for Improvement in Appearance of Gluteal Skin Irregularities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CASA2406
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Gluteal Skin Irregularities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Participants will receive three subcutaneous injection of single regimen of Sculptra 011611. A single regimen consists of up to three injection sessions spaced 1 month (+2 weeks) apart at Baseline, Month 1 and Month 2.
  Interventions: Device: Sculptra 016011
- Control Group (No Intervention): Participants will be randomized to not receive any intervention.

INTERVENTIONS:
Device: Sculptra 016011 — Freeze-dried powder for injection.
  Other Names: Poly L Lactic Acid (PLLA)
  Arms: Treatment Group

SUMMARY:
The main purpose of the study is to investigate the safety and effectiveness of Sculptra 011611 for improvement in appearance of gluteal skin irregularities.

ELIGIBILITY:
Inclusion Criteria:

* Participant with moderate to severe skin laxity in the buttocks when standing with the buttocks in repose as evaluated using the Buttocks' Skin Laxity Visual Scale (SLVS) by the Blinded Evaluator and Treating Investigator at the Baseline visit.
* Women 18 years of age and older.
* Has intent to undergo treatment to improve skin quality and skin irregularities in the buttock area.

Exclusion Criteria:

* Previous surgery in or near the treatment area.
* Previous treatment/procedure in or near the treatment area OR is planning to undergo any procedures affecting the treatment area, at any time during the study.
* Presence of any disease or lesions near or on the area to be treated.
* Evidence of scar-related disease or delayed healing activity within 1 year prior to the Baseline visit, or participants susceptible to keloid formation, hyperpigmentation or hypertrophic scarring from injectable procedures.
* Skin coloring/bleaching/tattoo/stretch marks in the treatment area, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
* An underlying known disease, a surgical or medical condition that would expose the participant to undue risk.
* Treatment with chemotherapy, immunosuppressive agents, topical and systemic prescription retinoids, topical and systemic corticosteroids within 3 months before treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders Having At Least "Improved" in Both Buttocks at Maximal Contraction According to the Global Aesthetic Improvement Scale (GAIS), as Assessed Live by Blinded Evaluator, at Month 9 | At Month 9
  Responder will be defined as participants achieving 'very much improved', 'much improved' or "Improved" on GAIS compared to baseline. The 7-graded GAIS will be used to assess the aesthetic improvement of gluteal skin irregularities by the Blinded Evaluator at maximal contraction by responding to the question: "How would you describe the aesthetic improvement today compared to the photograph taken at Baseline?" for each buttock separately by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse. In this outcome measure, percentage of participants who will achieve at least 'Improved' on the GAIS assessed by Blinded Evaluator at Month 9 will be reported.

SECONDARY OUTCOMES:
Percentage of Responders Having At Least "Improved" in Appearance of Gluteal Skin Irregularities in Both Buttocks at Maximal Contraction According to GAIS, as Assessed Live by Blinded Evaluator, at Month 3, 6 and 12 | At Months 3, 6 and 12
  Responder will be defined as participants achieving 'very much improved', 'much improved' or "Improved" on GAIS compared to baseline. The 7-graded GAIS will be used to assess the aesthetic improvement of gluteal skin irregularities by the Blinded Evaluator at maximal contraction by responding to the question: "How would you describe the aesthetic improvement today compared to the photograph taken at Baseline?" for each buttock separately by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse. In this outcome measure, percentage of participants who will achieve at least 'Improved' on the GAIS assessed by Blinded Evaluator at Months 3, 6 and 12 will be reported.
Percentage of Responders Having at Least "Improved" in Appearance of Gluteal Skin Irregularities in Both Buttocks in Relaxed State According to GAIS, as Assessed Live by Blinded Evaluator, at Month 3, 6, 9 and 12 | At Months 3, 6, 9 and 12
  Responder will be defined as participants achieving 'very much improved', 'much improved' or "Improved" on GAIS compared to baseline. The 7-graded GAIS will be used to assess the aesthetic improvement of gluteal skin irregularities by the Blinded Evaluator in relaxed state by responding to the question: "How would you describe the aesthetic improvement today compared to the photograph taken at Baseline?" for each buttock separately by using the respective categorical scale as follows; Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse. In this outcome measure, percentage of participants who will achieve at least 'Improved' on the GAIS assessed by Blinded Evaluator at Months 3, 6, 9 and 12 will be reported.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Site 8688, Vancouver, British Columbia
  - Site 7049, Vancouver, British Columbia
  - Site 8379, Burlington, Ontario
  - Site 8689, Toronto, Ontario
  - Site 8162, Woodbridge, Ontario
  - Site 8690, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: No